CLINICAL TRIAL: NCT00248222
Title: Early Aerobic Training Program After Ischemic Stroke
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Prof. David Tanne, Chaim Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-05-3840-DT-CTIL
Record Dates: First submitted 2005-11-02; First posted 2005-11-03 (Estimated); Last update posted 2009-10-27 (Estimated); Status verified 2009-10

CONDITIONS: Stroke; Cerebrovascular Accident
Keywords: Exercise; Rehabilitation; Aerobic training
MeSH Terms: conditions — Stroke; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Supervised aerobic training

SUMMARY:
The purpose of this study is to examine the feasibility and efficacy of an early supervised aerobic exercise program for patients following a minor ischemic stroke.

DETAILED DESCRIPTION:
The purpose of this study is to examine the feasibility and efficacy of an early supervised aerobic exercise program for patients following a minor ischemic stroke. Patients after a minor ischemic stroke would be randomized within 1-3 weeks of stroke onset to a control group (6 weeks of low intensity stretching and coordination exercises followed by a supervised aerobic training program) or an experimental group (immediate aerobic training program). Patients will be evaluated for measures of ambulation endurance, mobility, gait, functional assessment and clinical follow-up after 6 weeks and again 3 months later.

ELIGIBILITY:
Inclusion Criteria:

* minor ischemic stroke

Exclusion Criteria:

* unstable angina
* severe lung disease
* severe symptomatic peripheral vascular disease
* dementia or other severe neurological disease
* other severe uncontrolled medical problem

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-10; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
6 Minute Walk Test at 6 weeks
Modified Bruce Exercise Test at 6 weeks
Activity by Ankle accelerometer at 6 weeks

SECONDARY OUTCOMES:
Recurrent vascular events at 6 weeks
METS at 6 weeks
Stair climbing ascend and descend test at 6 weeks
Four Square Step Test at 6 weeks
Gait symmetry by SmartStep at 6 weeks
Walking Impairment Questionnaire at 6 weeks
Rivermead Mobility Index at 6 weeks
Similar outcome measures 3 months later

CONTACTS AND LOCATIONS:
Overall Officials: David Tanne, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Chaim Sheba Medical Center, Tel Litwinsky, Israel